CLINICAL TRIAL: NCT04657367
Title: Polish Registry of Diabetes - PL: Polski Rejestr Diabetologiczny (PolReD)
Brief Title: Polish Registry of Diabetes (PolReD)
Acronym: PolReD
Status: Recruiting | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Other Study IDs: R-I- 002/436/2019
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-11

CONDITIONS: Diabetes; Obesity; PreDiabetes; Dysglycemia
Keywords: diabetes registry; prediabetes registry
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Prediabetic State

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Diabetes: Patients with diagnosed diabetes
  Interventions: Other: Observational study - registry
- Prediabetes: Patients with diagnosed prediabetes defined as impaired fasting glucose and/or impaired glucose tolerance
  Interventions: Other: Observational study - registry
- Normoglycemia: Patients with normoglycemia, based on the OGTT - normal fasting glucose and normal glucose tolerance
  Interventions: Other: Observational study - registry

INTERVENTIONS:
Other: Observational study - registry — Observational study - registry

SUMMARY:
The aim of this project is to create a registry of diabetic patients, containing a detailed clinical profile of each patient, along with omics data, which will be analyzed using artificial intelligence algorithms, and their results will be implemented in the form of new recommendations of care for high-risk patients and those already suffering from diabetes.

The study will be conducted prospectively. The project participants will be patients with diabetes, patients at high risk of developing diabetes and a control group of normoglycemic patients who will participate in study visits at the Clinical Research Center of the Medical University of Bialystok.

DETAILED DESCRIPTION:
The aim of this project is to create a registry of patients at risk of developing diabetes or already diagnosed with diabetes, containing a detailed clinical profile of each patient, along with omics data, which will be analyzed using artificial intelligence algorithms, and their results will be implemented in the form of new recommendations of care for high-risk patients and those already suffering from diabetes.

The study will be conducted prospectively. The project participants will be patients with diabetes, patients at high risk of developing diabetes and a control group of normoglycemic patients who will participate in study visits at the Clinical Research Center of the Medical University of Bialystok.

As part of the project, each patient will participate in one visit at the research center. During the visit, each patient will undergo a detailed medical interview regarding the current health condition, the course of previously diagnosed diseases, family history, physical activity and diet. In addition, venous blood will be taken for each patient, from which the basic metabolic parameters will be determined (including glucose, lipid profile, HbA1c, AST, ALT, GGTP, electrolytes, blood count with smear, presence of antibodies against beta-cell antigens, TSH, ACTH) and omics analyzes will be performed (including genotyping and sequencing of DNA, transcriptomics, metabolomics, proteomics and lipidomics). Additionally, from each patient, saliva, urine, stool sample, and skin and nasal swabs to assess the microbiome will be collected. Each patient will also receive a detailed body composition analysis using bioimpedance and densitometry (DXA) and grip strength analysis. Non-diabetic patients will also undergo an oral glucose load test (OGTT).

In addition, patients who give additional consent will be able to participate in additional visits, including abdominal MR imaging with the assessment of liver steatosis, a biopsy of the vastus lateralis muscle, cardio-pulmonary exercise test, metabolic clamp (euglycemic - hyperinsulinemic) and glycemia assessment using the continuous glucose monitoring system ( CGM).

As part of the project, we plan for follow-up each participant with re-visits in the study centre every five years, covering exactly the same schedule of visits as the patient will make the first time.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosed diabetes (according to the American Diabetes Association criteria) - diabetes group
* patients with diagnosed prediabetes (IFG and/or IGT) - prediabetes group
* patients with normoglycemia (NFG and NGT) - normoglycemia group
* informed consent

Exclusion Criteria:

* drug addiction
* severe psychiatric disorders
* patients with gestational diabetes mellitus
* patients unable to give informed consent, legally incompetent or incapable to comply with the study terms and conditions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The project participants will be patients with diabetes, patients at high risk of developing diabetes (prediabetes) and a control group of normoglycemic patients from Poland.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | every 5 years
  Haemoglobin A1c measured by the high-performance liquid chromatography (HPLC) method
Fasting glucose | every 5 years
  Fasting glucose concentration measured in plasma using the colorimetric method
2-hour glucose | every 5 years
  Glucose concentration at 2-hour of the oral glucose tolerance test, measured in plasma using the colorimetric method - only in non-diabetic subjects
Fasting insulin | every 5 years
  Fasting insulin concentration measured in plasma using the immunoradiometric assay (IRMA)
Lean body mass | every 5 years
  Total lean body mass measured using the whole-body dual-energy X-ray absorptiometry (DXA)
Fat mass | every 5 years
  Total body fat mass measured using the whole-body dual-energy X-ray absorptiometry (DXA)
Visceral Adipose Tissue mass | every 5 years
  Visceral adipose tissue mass measured using the whole-body dual-energy X-ray absorptiometry (DXA)
Weight | every 5 years
  Total body weight measured using standardized scale
Homeostatic model assessment for insulin resistance (HOMA-IR) | every 5 years
  Homeostatic model assessment for insulin resistance
Homeostatic model assessment of beta cell function (HOMA-beta) | every 5 years
  Homeostatic model assessment of beta cell function
VO2max | every 5 years
  Maximal oxygen consumption measured during cardio-pulmonary exercise test
Triglycerides (TG) | every 5 years
  Serum triglycerides concentration measured using colorimetric method
High-density lipoprotein cholesterol (HDL) | every 5 years
  Serum high-density lipoprotein cholesterol (HDL) concentration measured using colorimetric method Serum high-density lipoprotein cholesterol (HDL) concentration measured using colorimetric method
  Serum high-density lipoprotein cholesterol (HDL) concentration measured using colorimetric meth
Low-density lipoprotein cholesterol (LDL) | every 5 years
  Serum low-density lipoprotein cholesterol (LDL) concentration measured using colorimetric method
Total cholesterol | every 5 years
  Serum total cholesterol concentration measured using colorimetric method
Plasma metabolome | every 5 years
  plasma metabolites concentrations measured using untargeted metabolomics
Skeletal muscle transcriptome | every 5 years
  skeletal muscle gene and smallRNA expressions measured using untargeted transcriptomics
Skeletal muscle metabolome | every 5 years
  skeletal muscle metabolites concentrations measured using untargeted metabolomics
Plasma microRNAs | every 5 years
  Expression of circulating smallRNA

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Centre, Medical University of Bialystok, Bialystok, Podlaskie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided